CLINICAL TRIAL: NCT02440074
Title: Lumbar Degenerative Disc Disease Treatment With Bone Marrow Autologous Mesenchymal Stem Cells (MSV)
Acronym: MSV-DISC
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Not funded Administrative formalities not completed
Sponsor: Red de Terapia Celular (Industry)
Collaborators: Instituto de Salud Carlos III (Other Government); University of Valladolid (Other); Centro en Red de Medicina Regenerativa de Castilla y Leon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eudra-CT2008-001191-68; MSV-DISC-2008-01 (Other Grant/Funding Number: Advenced Therapies Program, MICINN, Spain)
Record Dates: First submitted 2015-05-04; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Degenerative Disc Disease
Keywords: Lumbar pain; Mesenchymal Stem Cells
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain | interventions — Genes, mos

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSV autologous transplantation (Experimental)
  Interventions: Other: Autologous bone marrow mesenchymal stem cells

INTERVENTIONS:
Other: Autologous bone marrow mesenchymal stem cells — Bone marrow collection from patient, mesenchymal cells isolation and expansion under Good Manufacturing Practice (GMP) conditions following the IBGM-Valladolid protocol (MSV). Autologous MSV implantation by intradiscal injection.
  Other Names: MSV, mesenchymal stem cells by IBGM-Valladolid protocol.

SUMMARY:
This trial pretends to validate for clinical use a bioengineered product composed of mesenchymal stem cells produced by the Instituto de Biologia y Genetica Molecular (IBGM), Valladolid (MSV, which have already been approved by the Spanish Regulatory Agency for three previous clinical trials) and a cross-linked matrix of autologous plasma patented by The Blood and Tissue Bank of Asturias (WO2008/ 119855) for bone maxillary cysts refilling. These two groups collaborate in the present project with the team of Maxillofacial Surgery of the Hospital Universitario del Río Hortega, who leads the clinical trial and deals with the medical aspects. The proposed trial is based on positive results obtained in previous animal studies performed by the present multidisciplinary team. A phase I / II clinical trial with 10 patients suffering from bone cysts in the maxillofacial region is proposed. Autologous mesenchymal stem cells isolated from a bone marrow sample will be seeded in the autologous plasma matrix and cultivated for 3 weeks. At this time, the cyst will be removed by surgery and the cavity filled with the protein matrix containing the mesenchymal cells. Follow up tests will be conducted at 3 weeks, 3 and 6 months following the evolution of the cavity by panoramic radiography and computerized tomography scan.

DETAILED DESCRIPTION:
The proposed test is based on previous animal experiments with positive results by the multidisciplinary team applicant, whose results are presented in paragraph 2.6 (group results Valladolid) and Annex I (group results Oviedo).

The investigators propose phase I-II trial with 10 patients with a common condition and difficult to solve volumetric regeneration therapies, such as bone cysts in the maxillofacial region.

Autologous mesenchymal cells isolated from a sample obtained from the cancellous bone of the tuberosity intraoral mandibular later and after expansion, will be conveyed in the matrix of autologous serum. The total process takes 6-8 weeks. After this time, perform the osteotomy and enucleation of the cyst under local anesthesia and the residual cavity is filled with bioimplant containing the MSV-H.

Once the bioimplant, there will be clinical controls at 2 weeks, 2 and 6 months, to follow the evolution of regeneration by bone cavity in panoramic radiograph and CT scan.

This project proposes a novel approach to therapy twice, combining a tissue engineering protocol (bioimplant) consisting of autologous mesenchymal cells have already been approved by the unit cell production of Valladolid (MSV-H), and a new protein matrix obtained autologous serum crosslinked in order to stimulate the regenerative capacity of maxillary cystic bone defects.

ELIGIBILITY:
Inclusion Criteria:

* Degenerative disease of one or two lumbar discs with predominant back pain after conservative treatment (physical and medical) for over 6 months.
* Fibrous ring capable of holding the cell implantation, demonstrated by Magnetic Resonance Imaging (MRI; stages 2, 3 and 4 of Adams).
* Decrease of disc height of more than 20% (radiographic measurement in side image).
* Absence of spinal infection.
* Haematological and biochemical analysis wit no significant alterations that contraindicates intervention.
* The patient is able to understand the nature of the study.
* Informed written consent of the patient.

Exclusion Criteria:

* Age over 75 or under 18 or legally dependent
* Allergy to gentamicin, or to bovine, cattle or horse serum.
* Congenital or acquired diseases leading to spine deformations that may upset cell application.
* Spinal segmental instability, spinal canal stenosis, isthmus pathology and other conditions that may compromise the study
* Modic III changes on MRI images (31).
* Overweight with body mass index (mass in Kg/size in m2) greater than 35 (obesity grade II).
* Pregnancy or breast-feeding
* Neoplasia
* Immunosuppression
* Participation in another clinical trial or treatment with another investigational product within 30 days prior to inclusion in the study.
* Other conditions that may, according to medical criteria, discourage participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Pain relief | Change from baseline at 12 months after intervention.
  Pain is scored between 0 and 100 in Visual Analogue Scale for pain (VAS).